CLINICAL TRIAL: NCT01408784
Title: Evaluating the Validity of the "Categories" Method: a New Method for Self-report Assessment of Daily Calorie Intake
Brief Title: A New Method for Self-assessment of Daily Calorie Intake
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assuta Hospital Systems (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other); Rabin Medical Center (Other)
Responsible Party: Tzachi KNAAN, Maccabi health services
Other Study IDs: 172011
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2011-07

CONDITIONS: Diet Records; Caloric Restriction
Keywords: calories; counting; obesity; overweight; categories; calorie; method; counting calories; lose weight; diet; energy balance; energy intake; 24 hours recall; food intake
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the validity of self-caloric evaluation, the "categories method" - a new method based on one categorical score per meal

DETAILED DESCRIPTION:
Weight loss is mainly a result of reduction in daily caloric intake. Hence many people are interested in counting and tracking their daily caloric intake but In fact only 9% of people in the USA can accurately estimate the number of calories they eat (International Food Information Council Foundation, May 2011)

According to the well-known method the investigators need to know the caloric value of each and every component our dish or meal. For example: a Breakfast that contains a glass of orange juice, a small bagel, spread with cream cheese shall be calculated as : orange juice 90 kcal + bagel 192 kcal +cream cheese 98 kcal=total 380 kcal.

This method is very complicated, especially when the investigators need to calculate a dish that its ingredients are not straightforward such as: Cob salad or Shepherd's pie, Even a slice of pizza, it is very difficult to estimate the fat, carbohydrate or protein a piece of pie contains let alone the caloric volume.

The investigators proposed a new method called "The categories method": a single categorical estimation per meal based on a set of five categories:

Category 1 less than 200 kcal, Category 2 200-500 kcal, Category 3 501-800 kcal, Category 4 801-1200 kcal, Category 5 above 1200 kcal

After choosing the category the investigators use an average of the category (e.g., category 3: 500-800 Avg = 650 kcal). Using the same Breakfast description as above: this meal will be considered as category No. 2 (200-500 Kcal), and chicken and rice at the restaurant will considered as a category 4 (800-1200 Kcal).

This method simplifies the process of counting calories, especially with assembled or cooked meal, it makes it easier to track any given meal even to those how are not so familiar with the caloric value of a product.

Research protocol:Participates will interviewed face to face on 1 occasion to obtain 24 hours recall using 4 pass method include 1. Quick review of the meals. 2. Food items that may be forgotten 3. Time and place of each meal 4. Assessment of food quantities and dimensions using a photograph published by the Israeli Ministry

This method is implemented with U.S. Department of Agriculture (USDA) as part of nutritional surveys and is used for "MBT" Survey of the Israeli Ministry of Health

Using "Tzameret" software system (food composition program of the Israeli Ministry of Health) The investigators will input the 24HR recall food list and quantity to calculate caloric values for every meal and the total calorie intake.

Using the "Categories Method" the investigators will calculate the caloric value of a meal by giving the average value of each category (record in parentheses).

Finally, reliability of the "categories method" compare with the 24HR recall will statistically calculated.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-65
* Body mass index (BMI) between 20-45 kg/m2
* Workers of Maccabi Healthcare Services
* Members of Maccabi Healthcare Services

Exclusion Criteria:

-Clinical dietitians / Nutritionists

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Total Calorie intake using "categories method" | 30-45 minutes
  Sum of every meal (the average)

SECONDARY OUTCOMES:
Total calories per meal using "categories method" | 30-45 minutes
  Average of a category

CONTACTS AND LOCATIONS:
Overall Officials: Orit Klinger, MD, Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- Maccabi Healthcare Services, Tel Aviv, Israel